CLINICAL TRIAL: NCT01142609
Title: Improving Substance Abuse Counseling Adherence Using Web-based Videoconferencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Van King, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1RC1DA028189-01 (NIH); 1RC1DA028189-01 (NIH)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Substance Abuse Disorder
Keywords: Web based videoconferencing; methadone; substance abuse counseling
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet (eGetgoing) (Experimental): Subjects will assigned to use an accredited web-based platform (eGetgoingTM, CRC Health Group, Inc.) to deliver routine substance abuse counseling.
  Interventions: Behavioral: eGet
- Routine on-site (No Intervention): Subjects will attend routine face-to-face individual counseling sessions.

INTERVENTIONS:
Behavioral: eGet — eGet individual counseling sessions from home will be scheduled weekly for 12 weeks.
  Arms: Internet (eGetgoing)

SUMMARY:
This research is being done to compare the effectiveness of standard on-site, in-person counseling with Internet web-based videoconferencing (e-therapy) in drug-dependent patients in opioid-agonist treatment programs. The study is looking to see if there are any differences in satisfaction or in treatment outcome if counseling sessions are given by e-therapy compared to standard, in-person counseling given in the clinic. The e-therapy happens in real time- it works very much like standard therapy in the clinic except that the patient is in his or her own home (or other convenient location outside the clinic) and talks to and sees the therapist through an Internet connection on the computer (the therapist will usually be at the clinic).

DETAILED DESCRIPTION:
This study will be the first to evaluate the efficacy of an accredited and currently available, Internet web-based videoconferencing platform to deliver routine schedules of counseling in an opioid agonist treatment program. It has outstanding potential to help determine transportability of this technology to other treatment programs by demonstrating the benefits of integration of web-based therapy with on-site services to expand the continuum of care.

ELIGIBILITY:
Inclusion Criteria:

* Access to a computer with Internet capability
* Full adherence to their routine counseling schedule over the previous 30-days
* Negative urine specimens over the previous 30-days
* Patient at ATS for 90 days

Exclusion Criteria:

* No access to a computer with Internet capability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Counseling efficacy | Weekly for 12 weeks
  Attendance to individual counseling sessions, both online and on-site will be tracked weekly for the duration of the study.
Reinforcement value (eGetgoing) | Monthly for 3 months
  Subjects will complete monthly surveys to evaluate the reinforcement value of eGetgoing using a multiple choice design that will compare its perceived value to other aspects of routine treatment (e.g., take-home medications).
Reinforcement value (on-site) | Baseline
  Subjects will complete a survey to evaluate the reinforcement value of eGetgoing using a multiple choice design that will compare its perceived value to other aspects of routine treatment (e.g., take-home medications).

SECONDARY OUTCOMES:
Program Satisfaction | Baseline and monthly for 3 months
  Subjects will complete a survey to assess their overall program satisfaction
Treatment cost | Baseline and Month 3
  Subjects will complete surveys to measure treatment related time and monetary travel costs.
Therapeutic relationship | Baseline and monthly for 3 months
  Subjects and their therapists will complete surveys to assess qualities of the therapeutic relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Van King, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services, Baltimore, Maryland, United States